CLINICAL TRIAL: NCT03332459
Title: A Long-term Follow-up of Study 64041575RSV2004 to Evaluate the Impact of Lumicitabine (JNJ-64041575) on the Incidence of Asthma and/or Wheezing in Infants and Children With a History of Respiratory Syncytial Virus Infection
Brief Title: A Long-term Follow-up Study to Evaluate the Impact of Lumicitabine on the Incidence of Asthma and/or Wheezing in Infants and Children With a History of Respiratory Syncytial Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108375; 2016-002095-26 (EudraCT Number); 64041575RSV2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumicitabine (Experimental): Participants who completed the last planned study-related visit in a feeding Phase 2 study (64041575RSV2004), in which they received a regimen containing lumicitabine for the treatment of RSV infection, and who agree to participate in this follow-up study will be assessed for the incidence of the clinical diagnosis of asthma, frequency of wheezing, long-term safety of lumicitabine, frequency and type of respiratory infections and medical resource usage.
  Interventions: Drug: Lumicitabine
- Placebo (Placebo Comparator): Participants who completed the last planned study-related visit in a feeding Phase 2 study (64041575RSV2004), in which they received a regimen containing placebo for the treatment of RSV infection, and who agree to participate in this follow-up study will be assessed for the incidence of the clinical diagnosis of asthma, frequency of wheezing, long-term safety of placebo, frequency and type of respiratory infections and medical resource usage.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumicitabine — Participants who received lumicitabine in a feeding Phase 2 study (64041575RSV2004) will be observed in this study.
  Arms: Lumicitabine
Drug: Placebo — Participants who received placebo in a feeding Phase 2 study (64041575RSV2004) will be observed in this study.
  Arms: Placebo

SUMMARY:
The purpose of this long-term follow-up (LTFU) study is to evaluate the incidence of the clinical diagnosis of asthma and the frequency of wheezing in infants and children with respiratory syncytial virus (RSV) infection who were treated with (lumicitabine or placebo) and have completed their last planned study-related visit in a feeding Phase 2 study (64041575RSV2004).

DETAILED DESCRIPTION:
RSV is a leading cause of lower respiratory tract disease in infants. The primary hypothesis is that treatment of RSV-infected infants/children with lumicitabine (also known as JNJ-64041575 or ALS-008176) will decrease subsequent wheezing/asthma compared to placebo (looks like lumicitabine). The participants who have completed treatment course (lumicitabine/placebo) and last study visit in a previous study, 64041575RSV2004, for the treatment of RSV infection will be enrolled in this LTFU study. The main purpose of this study is to understand the impact of lumicitabine on the occurrence of asthma/wheezing in infants/children with a history of RSV infection. The participants will be assessed via monthly calls with the parents/caregivers and also at site visits at 3, 6,12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants and children who were previously randomized in study 64041575RSV2004 for the treatment of respiratory syncytial virus (RSV) infection and who completed the planned course of the study drug and the last study-related visit of study 64041575RSV2004
* The participant's legally acceptable representative must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing for the participant to participate in the study

Exclusion Criteria:

* The participants legally acceptable representative, i.e, parent/legal guardian/caregiver, is not able to maintain reliable communication with the investigator
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Ages: 56 Days to 39 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- Japan (4):
  - Fukuyama City Hospital, Fukuyama
  - Hirosaki National Hospital, Hirosaki
  - National Hospital Organization Niigata National Hospital, Niigata
  - National Hospital Organization Beppu Medical Center, Ōita

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who previously received lumicitabine or placebo in study 64041575RSV2004 (NCT03333317) were enrolled in this long term follow-up (LTFU) study.
Groups:
- Placebo: Participants who had received placebo for the treatment of respiratory syncytial virus (RSV) infection during study 64041575RSV2004 and continued to participate in this long term follow-up (LTFU) study were assessed for the clinical diagnosis of asthma and wheezing in infants and children.
- Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD): Participants who had received lumicitabine 40 mg/kg as LD (Dose 1) followed by 9 MD doses of lumicitabine 20 mg/kg twice a day for the treatment of RSV infection during study 64041575RSV2004 and continued to participate in this LTFU study were assessed for the clinical diagnosis of asthma and wheezing in infants and children.
- Lumicitabine 60/40 mg/kg LD/MD: Participants who had received lumicitabine 60 mg/kg as LD (Dose 1) followed by 9 MD doses of lumicitabine 40 mg/kg twice a day for the treatment of RSV infection during study 64041575RSV2004 and continued to participate in this LTFU study were assessed for the clinical diagnosis of asthma and wheezing in infants and children.
Period: Overall Study
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Started | 3 | 1 | 3
Completed | 3 | 1 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD | Total
Number analyzed (Participants) | 3 | 1 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: months] | 16 (13.08) | 17 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 6.3 (2.52) | 12 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 3 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 2 | 5
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  JAPAN | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Asthma After Respiratory Syncytial Virus (RSV) Infection
Description: Percentage of participants with asthma diagnosed by physician were reported.
Time Frame: Up to 2 years
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this long term follow up (LTFU) study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
percentage of participants | 0 [0 to 56.15] | 0 [0 to 79.35] | 0 [0 to 56.15]

2. Primary Outcome: Percentage of Wheezing Days in Participants Within the First 2 Years After RSV Infection
Description: Percentage of wheezing days in participants within the first 2 Years after RSV infection based on information reported by the parent/caregiver were reported. Percentage of wheezing days was calculated by (number of wheezing days/days of study completion - day of informed consent + 1)*100.
Time Frame: Up to 2 years
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this LTFU study.
Measure: Mean (Standard Deviation); unit: percentage of wheezing days
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
percentage of wheezing days | 0.03 (0.058) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 2.53 (4.388)

3. Secondary Outcome: Percentage of Wheezing Days in Participants Per Month After RSV Infection
Description: Percentage of wheezing days in participants per month after RSV infection based on information reported by the parent/caregiver were reported. Percentage of wheezing days per month was calculated by number of days reported in that period with wheezing, using last day - first day + 1 for reported days of wheezing and multiplied by 100%.
Time Frame: Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this LTFU study.
Measure: Mean (Standard Deviation); unit: percentage of wheezing days per month
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
percentage of wheezing days per month
  Month 1 | 1.00 (1.732) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 1.00 (1.732)
  Month 2 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 1.00 (1.732)
  Month 3 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 5.67 (9.815)
  Month 4 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 5 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 6 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 2.00 (3.464)
  Month 7 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 8 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 9 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 4.33 (7.506)
  Month 10 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 3.33 (5.774)
  Month 11 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 5.00 (8.660)
  Month 12 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 5.67 (9.815)
  Month 13 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 6.33 (10.970)
  Month 14 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 4.33 (7.506)
  Month 15 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 6.00 (10.392)
  Month 16 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 7.67 (13.279)
  Month 17 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 4.00 (6.928)
  Month 18 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 19 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 20 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 1.00 (1.732)
  Month 21 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 22 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 23 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 4.00 (6.928)
  Month 24 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)

4. Secondary Outcome: Number of Wheezing Episodes in Participants Per Month After the RSV Infection
Description: Number of wheezing episodes in participants per month after the RSV infection based on information reported by the parent/caregiver were reported.
Time Frame: Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this LTFU study.
Measure: Mean (Standard Deviation); unit: wheezing episodes per month
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
wheezing episodes per month
  Month 1 | 0.33 (0.577) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 2 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 3 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 4 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 5 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 6 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 7 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 8 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 9 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 10 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 11 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 1.00 (1.732)
  Month 12 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 1.00 (1.732)
  Month 13 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 1.00 (1.732)
  Month 14 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.67 (1.155)
  Month 15 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 16 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 17 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 18 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 19 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 20 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.33 (0.577)
  Month 21 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 22 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)
  Month 23 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.67 (1.155)
  Month 24 | 0.00 (0.00) | 0.00 (NA) — Here 'NA' signifies that standard deviation was not calculated as only one participant was evaluated. | 0.00 (0.00)

5. Secondary Outcome: Number of Participants With Reportable Adverse Events (AEs)
Description: Number of participants with reportable AEs were reported. The following AEs were considered reportable (within the context of this study): respiratory illness AEs, including subsequent RSV infections, adverse events considered at least possibly related to study treatment (lumicitabine or placebo, as received in study 64041575RSV2004), and serious adverse events.
Time Frame: Up to 2 years
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this LTFU study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 3 | 1 | 2

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 2 years
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this LTFU study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants | 0 | 0 | 1

7. Secondary Outcome: Number of Respiratory Infections Per Participant
Description: The number of respiratory infections per participant, based on information reported by the parent/caregiver were reported.
Time Frame: Up to 2 years
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this LTFU study. Here 'N' (number of participants analyzed) included all participants who had a respiratory infection.
Measure: Mean (Standard Deviation); unit: infections per participant
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 2
infections per participant | 10.7 (4.62) | 6.0 (0.00) | 19.5 (6.36)

8. Secondary Outcome: Number of Participants With Medical Encounters
Description: Number of participants with medical encounters (hospital inpatient department visits, hospital outpatient department visits, medical practitioner office visits) was reported based on information reported by the parent/caregiver.
Time Frame: Up to 2 years
Population: All Enrolled analysis set included all participants from 64041575RSV2004 study who were enrolled in this LTFU study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
Number analyzed (Participants) | 3 | 1 | 3
Participants
  Hospital Inpatient Department Visits | 0 | 0 | 1
  Hospital Outpatient Department Visits | 3 | 1 | 2
  Medical Practitioner Office Visits | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 2 years (during this long term follow up study)
Description: Reportable AEs (Respiratory illness AEs, including subsequent RSV infections, AEs considered at least possibly related to study treatment [lumicitabine or placebo, as received in Study 64041575RSV2004], and serious adverse events) reported below. All Enrolled analysis set: all participants from 64041575RSV2004 study enrolled in this LTFU study.
Arm/Group | Placebo | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) | Lumicitabine 60/40 mg/kg LD/MD
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) (N=1) | Lumicitabine 60/40 mg/kg LD/MD (N=3)
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1
Exanthema Subitum (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Norovirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Rotavirus (Infections and infestations) | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Lumicitabine 40/20 Milligrams/Kilogram (mg/kg) Loading Dose/Maintenance Dose (LD/MD) (N=1) | Lumicitabine 60/40 mg/kg LD/MD (N=3)
Adenovirus Infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1
Enterocolitis Viral (Infections and infestations) | 0 | 0 | 1
Exanthema Subitum (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the limited number of participants enrolled in this study (n=7), no meaningful conclusions can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT03332459/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT03332459/SAP_001.pdf